CLINICAL TRIAL: NCT05054699
Title: Electroconvulsive Therapy Versus Magnetic Seizure Therapy: Clinical and Cognitive Outcomes
Brief Title: Electro-Magnetic Convulsive Therapies for Depression: a Non-inferiority Study
Acronym: EMCODE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Andre R Brunoni, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29979220.4.0000.0068
Record Dates: First submitted 2021-09-05; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder; Bipolar Depression
Keywords: Magnetic Seizure Therapy; Electroconvulsive Therapy; Depression; Major Depressive Disorder; Bipolar Depression; Cognition
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly and blindly allocated to either of two interventions, namely, MST or ECT. Clinical and cognitive parameters will be assessedat baseline, weeks 6, 12 and 18.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be anaesthetised before the procedure, therefore will not be able to tell whether they received ECT ou MST. The preparation procedures before seizure will be identical for all participants regardless of the intervention. All monitoring and other procedures will be exactly the same for both groups. Investigator and rater will not have access to which procedure subjects received. To blind the staff, the MST sound will performed during all study interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- MST (Experimental): Subjects will receive 12-18 sessions of frontal Magnetic Seizure Therapy under general anaesthesia, twice a week. Clinical and cognitive measures will be assessed before, during and after the treatment
  Interventions: Device: Magnetic Seizure Therapy
- ECT (Active Comparator): Subjects will receive 12-18 sessions of bilateral Electroconvulsive Therapy under general anaesthesia, twice a week. Clinical and cognitive measures will be assessed before, during and after the treatment
  Interventions: Device: Electroconvulsive Therapy

INTERVENTIONS:
Device: Magnetic Seizure Therapy — Subjects will receive a train of magnetic pulses (between 600 and 1400 pulses) at 100Hz under general anaesthesia using a Magventure device with a Twin Coil
  Other Names: MST
  Arms: MST
Device: Electroconvulsive Therapy — Subjects will receive a brief-pulse electrical stimulus (between 25 and 1008mC) under general anaesthesia using a ECT device
  Other Names: ECT
  Arms: ECT

SUMMARY:
This study aims to compare the efficacy and safety profile of Magnetic Seizure Therapy and Electroconvulsive therapy.

DETAILED DESCRIPTION:
Magnetic seizure therapy (MST) is a novel, experimental therapeutic intervention, which combines therapeutic aspects of electroconvulsive therapy (ECT) and transcranial magnetic stimulation, in order to achieve the efficacy of the former with the safety of the latter. While ECT remains the most efficacious treatment available for severe and treatment-resistant depression, it is hampered by its side effect profile, specially cognitive deficits, which albeit transitory might be particularly distressing for patient, not to mention the stigma that still clings to this method. MST employs high frequency magnetic pulses applied to the head to the patient in order to induce generalized epileptic activity, thus emulating the core feature of ECT. Though distributed over a large area, such pulses do not penetrate deeper areas of the brain, therefore sparing deeper areas such as the hippocampi, which are crucial for memory encoding.

The goal of this study is to compare the antidepressant action of MST to ECT, using a non-inferiority approach. It also aims to compare the cognitive side effects profile of both interventions, as well as investigate possible neuroimaging changes and response predictors before and after treatments.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder or Bipolar Depression in accordance to the Diagnostic and Statistical Manual (DSM) criteria
* Score equal to or great than 17 points on the Hamilton Depression Rating Scale
* Treatment-resistant depression, defined as insufficient relief of symptoms after two different first line treatments using therapeutic doses and for four to six weeks
* Adequate health and clinical conditions, as assessed by an anaesthesiologist and a psychiatrist

Exclusion Criteria:

* Pregnancy
* Other psychiatric conditions such as Schizophrenia, Schizoaffective Disorder, Substance Abuse, Borderline Personality Disorder, PTSD, or Intellectual Deficiency
* Depressive symptoms due to a clinical condition
* Any clinical or neurological conditions without proper management
* ECT or any other neuromodulation treatment on the last six months
* Inability to consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | Change from baseline to endpoint (week 18). However, the endpoint can be at week 12 if the patient is remitted at this time period.
  Score on the 17 items Hamilton Depression Rating Scale (HDRS-17). It measures the severity of clinical symptoms, ranging from 0 to 52, with higher scores indicating greater severity.
Biographical memory | Change from baseline to endpoint (week 18). However, the endpoint can be at week 12 if the patient is remitted at this time period.
  Score on the Autobiographical Memory Inventory (AMI). Interviewer-rated measure with 10 items that indexes autobiographical memory recall and specificity.

SECONDARY OUTCOMES:
Depressive Symptoms | Change from baseline to endpoint (week 18). However, the endpoint can be at week 12 if the patient is remitted at this time period.
  Score on the Montgomery-Asberg Depression Rating Scale (MADRS). It measures the severity of clinical symptoms, ranging from 0 to 60, with higher scores indicating greater severity.
Depressive Symptoms | Change from baseline to endpoint (week 18). However, the endpoint can be at week 12 if the patient is remitted at this time period.
  Score on the Beck Depression Inventory (BDI). It measures the severity of clinical symptoms, ranging from 0 to 63, with higher scores indicating greater severity.
Suicidal Thoughts | Change from baseline to endpoint (week 18). However, the endpoint can be at week 12 if the patient is remitted at this time period.
  Score on the Beck Scale for Suicidal Ideation (BSS). The BSS contains 19 items that measure the severity of actual suicidal wishes and plans. Scores range from 0 to 38, a higher score indicating a higher level of suicide ideation.

CONTACTS AND LOCATIONS:
Overall Officials: ANDRE R BRUNONI, Principal Investigator — FACULDADE DE MEDICINA DA USP
Locations (1):
- Institute of Psychiatry, HC-FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cretaz E, Bellini H, Gallucci-Neto J, Carneiro AM, Dos Santos LA, Miranda CS, Brunoni AR. Use of Magnetic Seizure Therapy for Treatment-Resistant Depression: A Case Series. J ECT. 2022 Dec 1;38(4):261-262. doi: 10.1097/YCT.0000000000000868. Epub 2022 Jul 19. No abstract available. PMID 35900079